CLINICAL TRIAL: NCT07117045
Title: Artificial Intelligence-powered Low-Dose Computed Tomography for Screening of Pancreatic Cancer
Acronym: AI-LDCT-PC
Status: Recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: Ningbo University Affiliated People's Hospital (Unknown); Jiaxing University Affiliated Second Hospital (Unknown); Meinian Onehealth Healthcare Holdings Co., Ltd (Unknown); Ruici Medical Examination Institution (Unknown)
Responsible Party: Sponsor
Other Study IDs: AI-LDCT-PC; 202401063 (Other Grant/Funding Number: Shanghai Municipal Bureau of Data); 202440208 (Other Grant/Funding Number: Shanghai Municipal Health Commission); 2025AAA031146 (Other Grant/Funding Number: National Science and Technology Major Project)
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Cancer; Intraductal Papillary Mucinous Neoplasm; High-grade Pancreatic Intraepithelial Neoplasia; PDAC - Pancreatic Ductal Adenocarcinoma; Mucinous Cystic Neoplasm
Keywords: Screening; Early Diagnosis; Pancreatic Cancer; Artificial Intelligence; Computed Tomography
MeSH Terms: conditions — Pancreatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will have the option to donate blood samples for biobanking. Approximately 20ml blood and 2ml serum will be collected. Additional samples collected for diagnostic purposes may be banked. If consented, biological samples (blood, tissue, saliva) will be used for identifying potential biomarkers from de-identified samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AI-powered LDCT (LDCT+AI): Participants will undergo annual screening with the LDCT+AI system.
  Interventions: Diagnostic Test: Diagnostic Evaluation for Positive AI Findings

INTERVENTIONS:
Diagnostic Test: Diagnostic Evaluation for Positive AI Findings — MDT will review positive AI findings (including PDAC, pancreatic precursor lesions and benign lesion) cases to determine next steps: (1) Suspected PDAC and pancreatic precursor lesions are referred for hospital examination with diagnostic results collected; (2) Benign lesion cases receive personalized monitoring until endpoint events or study end; (3) Cases with positive AI findings but MDT-confirmed normal pancreatic issues receive at least one year of follow-up. If any abnormal results arise, management will transition to either plan (1) or (2).

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) has a poor prognosis, with early diagnosis crucial for improving survival. Due to the absence of effective screening methods, most patients are diagnosed at advanced stages. The population undergoing low-dose computed tomography (LDCT) screening significantly overlaps with those at high risk for PDAC; however, traditional imaging methods have limited sensitivity for detecting pancreatic lesions. This study utilizes the Pancreatic Cancer Detection with Artificial Intelligence (PANDA) system to enhance LDCT for pancreatic cancer screening in a prospective, multicenter, observational cohort. PANDA will analyze LDCT images, followed by a multidisciplinary team (MDT) reassessment of abnormal interpretations. Based on MDT evaluation, individuals will be recalled for further examination, placed under a personalized follow-up plan, or monitored for at least one year. The primary outcomes include pancreatic cancer detection rate, positive predictive value, consensus rate, and recall rate, while secondary outcomes focus on early-stage cancers, resectable tumors, and safety indicators such as false positive rates and unnecessary procedures. This study aims to assess the effectiveness and safety of AI-assisted LDCT for PDAC detection, providing a practical solution for improving public health and enhancing early diagnostic capabilities.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) is an extremely aggressive cancer with a dismal 5-year survival rate of just 13%. The key to improving outcomes lies in early detection, as patients diagnosed at an early stage (IA) can achieve an 80% 5-year survival. However, current screening methods are limited, focusing only on high-risk populations and lacking effectiveness for the general public due to the cancer's relatively low incidence and high false-positive risks.

Contrast-enhanced CT (CE-CT), the primary imaging modality, faces barriers for widespread implementation due to its invasiveness, high costs, and need for contrast agents. In this context, low-dose CT (LDCT) emerges as a promising alternative, having demonstrated success in lung cancer screening by reducing radiation exposure. Retrospective analysis revealed that one-third of pancreatic abnormalities were missed during routine LDCT interpretations, suggesting the untapped potential of LDCT-based pancreatic lesion screening.

Breakthroughs in AI have transformed medical imaging. Our PANDA (pancreatic cancer detection with artifcial intelligence) system excels at pancreatic cancer detection, utilizing innovative registration techniques and a cascaded deep learning framework (UNet+Max-Deeplab) for comprehensive lesion analysis. Validated across 10 centers (6,239 patients), PANDA outperformed radiologists. Real-world testing (20,530 cases) demonstrated remarkable accuracy: 92.9% sensitivity and 99.9% specificity, maintaining 92.2% sensitivity even for small T1 tumors. On LDCT, PANDA achieved 0.979 AUC without protocol modifications, confirming "LDCT+AI" as a viable screening approach.

China's health check-up environment presents three key advantages: First, LDCT delivers just 1/4-1/5 the radiation of standard abdominal CT, staying within ICRP safety guidelines (<3mSv). Second, LDCT offers superior cost-effectiveness compared to CE-CT by eliminating contrast agent expenses. Third, China's extensive annual health check-up infrastructure provides an unparalleled foundation for widespread implementation.

In the study, we will conduct a prospective, multicenter, observational cohort design targeting a health check-up population, utilizing the PANDA system to enhance LDCT for pancreatic cancer screening. Initially, PANDA analyzes the LDCT images of participants and provides interpretation results. Subsequently, a multidisciplinary team (MDT) will re-evaluate the cases with positive AI findings (including PDAC, pancreatic precursor lesions and benign lesion) and determine whether to recall the individuals: (1) Suspected PDAC and pancreatic precursor lesions are referred for hospital examination with diagnostic results collected; (2) Benign lesion cases receive personalized monitoring until endpoint events or study end; (3) Cases with positive AI findings but MDT-confirmed normal pancreatic issues receive at least one year of follow-up. If any abnormal results arise, management will transition to either plan (1) or (2). The primary outcome measures include pancreatic cancer detection rate, positive predictive value, consensus rate, and recall rate. Secondary outcome measures include the proportion of early-stage pancreatic cancers and resectable tumors. Safety indicators include the false positive rate, the proportion of unnecessary invasive procedures, and the proportion of unnecessary surgeries.

This study aims to evaluate the effectiveness and safety of AI-powered LDCT in detecting pancreatic cancer within a health check-up population, offering a practical solution to improve public health and early diagnosis for pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 years and above.
2. Voluntary signing of informed consent.
3. Completion of LDCT examination.

Exclusion Criteria:

1. Previous history of pancreatic cancer.
2. Abdominal inflammation or diagnosis of acute pancreatitis within 6 months.
3. Poor image quality due to ascites, pancreatic trauma, thoracic/abdominal surgery, radiotherapy or chemotherapy.
4. Research subjects unable to complete follow-up due to physical or other reasons.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes asymptomatic individuals aged 50 years and above who have undergone routine low-dose chest CT (LDCT) scans at health check-up centers. Eligible participants must provide written informed consent and be willing to attend all scheduled follow-up visits. Exclusion criteria include a previous history of pancreatic cancer, abdominal inflammation or diagnosis of acute pancreatitis within 6 months, poor image quality due to ascites, pancreatic trauma, thoracic/abdominal surgery, radiotherapy or chemotherapy, and research subjects unable to complete follow-up due to physical or other reasons.
Sampling Method: Non-Probability Sample
Enrollment: 400000 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2030-12-30 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Pancreatic cancer detection rate | 2 years
  The proportion of individuals with abnormal AI assessment confirmed as pancreatic cancer or precancerous lesions among the total screened population
Positive predictive value | 2 years
  The proportion of individuals with abnormal AI assessment confirmed as pancreatic cancer or precancerous lesions among all individuals with abnormal AI assessment
Consensus rate | 2 years
  The proportion of individuals with abnormal AI assessment deemed suspicious for pancreatic cancer or precancerous lesions by MDT requiring recall among the total screened population.
Recall rate | 2 years
  The proportion of individuals actually recalled among the total screened population.

SECONDARY OUTCOMES:
Early-stage pancreatic cancer proportion | 2 years
  The proportion of individuals with abnormal AI assessment confirmed as early-stage pancreatic cancer among the total number of confirmed pancreatic cancer cases.
Resectable pancreatic cancer proportion | 2 years
  The proportion of individuals with surgically resectable pancreatic cancer among the total number of confirmed pancreatic cancer cases.

OTHER OUTCOMES:
False positive rate | 2 years
  The proportion of individuals with abnormal AI assessment who actually have benign conditions or no lesions, among the total number of individuals with abnormal AI assessment.
Unnecessary invasive examination proportion | 2 years
  The proportion of individuals with abnormal AI assessment who underwent invasive examinations but were found to have benign conditions or no lesions, among the total number of individuals with abnormal AI assessment.
Unnecessary surgery proportion | 2 years
  The proportion of individuals with abnormal AI assessment who underwent surgery but were confirmed to have benign lesions by postoperative pathology, among the total number of individuals with abnormal AI assessment.
Pancreatic cancer 5-year survival rate | 7 years
  The proportion of pancreatic cancer patients detected by AI who are still alive after 5 years of follow-up, among the total number of pancreatic cancer patients detected by AI.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Meinian Onehealth Healthcare Holdings Co., Ltd, Shanghai, Shanghai Municipality
  - Ruici Medical Examination Institution, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Jiaxing University Affiliated Second Hospital, Jiaxing, Zhejiang
  - Ningbo University Affiliated People's Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao K, Xia Y, Yao J, Han X, Lambert L, Zhang T, Tang W, Jin G, Jiang H, Fang X, Nogues I, Li X, Guo W, Wang Y, Fang W, Qiu M, Hou Y, Kovarnik T, Vocka M, Lu Y, Chen Y, Chen X, Liu Z, Zhou J, Xie C, Zhang R, Lu H, Hager GD, Yuille AL, Lu L, Shao C, Shi Y, Zhang Q, Liang T, Zhang L, Lu J. Large-scale pancreatic cancer detection via non-contrast CT and deep learning. Nat Med. 2023 Dec;29(12):3033-3043. doi: 10.1038/s41591-023-02640-w. Epub 2023 Nov 20. PMID 37985692
- [Background] Mizrahi JD, Surana R, Valle JW, Shroff RT. Pancreatic cancer. Lancet. 2020 Jun 27;395(10242):2008-2020. doi: 10.1016/S0140-6736(20)30974-0. PMID 32593337
- [Background] Pereira SP, Oldfield L, Ney A, Hart PA, Keane MG, Pandol SJ, Li D, Greenhalf W, Jeon CY, Koay EJ, Almario CV, Halloran C, Lennon AM, Costello E. Early detection of pancreatic cancer. Lancet Gastroenterol Hepatol. 2020 Jul;5(7):698-710. doi: 10.1016/S2468-1253(19)30416-9. Epub 2020 Mar 2. PMID 32135127
- [Background] Attiyeh MA, Chakraborty J, Doussot A, Langdon-Embry L, Mainarich S, Gonen M, Balachandran VP, D'Angelica MI, DeMatteo RP, Jarnagin WR, Kingham TP, Allen PJ, Simpson AL, Do RK. Survival Prediction in Pancreatic Ductal Adenocarcinoma by Quantitative Computed Tomography Image Analysis. Ann Surg Oncol. 2018 Apr;25(4):1034-1042. doi: 10.1245/s10434-017-6323-3. Epub 2018 Jan 29. PMID 29380093
- [Background] Ardila D, Kiraly AP, Bharadwaj S, Choi B, Reicher JJ, Peng L, Tse D, Etemadi M, Ye W, Corrado G, Naidich DP, Shetty S. End-to-end lung cancer screening with three-dimensional deep learning on low-dose chest computed tomography. Nat Med. 2019 Jun;25(6):954-961. doi: 10.1038/s41591-019-0447-x. Epub 2019 May 20. PMID 31110349
- [Background] Wood LD, Canto MI, Jaffee EM, Simeone DM. Pancreatic Cancer: Pathogenesis, Screening, Diagnosis, and Treatment. Gastroenterology. 2022 Aug;163(2):386-402.e1. doi: 10.1053/j.gastro.2022.03.056. Epub 2022 Apr 7. PMID 35398344
- [Background] Singhi AD, Koay EJ, Chari ST, Maitra A. Early Detection of Pancreatic Cancer: Opportunities and Challenges. Gastroenterology. 2019 May;156(7):2024-2040. doi: 10.1053/j.gastro.2019.01.259. Epub 2019 Feb 2. PMID 30721664
- [Background] Chu LC, Park S, Kawamoto S, Wang Y, Zhou Y, Shen W, Zhu Z, Xia Y, Xie L, Liu F, Yu Q, Fouladi DF, Shayesteh S, Zinreich E, Graves JS, Horton KM, Yuille AL, Hruban RH, Kinzler KW, Vogelstein B, Fishman EK. Application of Deep Learning to Pancreatic Cancer Detection: Lessons Learned From Our Initial Experience. J Am Coll Radiol. 2019 Sep;16(9 Pt B):1338-1342. doi: 10.1016/j.jacr.2019.05.034. No abstract available. PMID 31492412
- [Background] Gros L, Yip R, Zhu Y, Li P, Paksashvili N, Sun Q, Yankelevitz DF, Henschke CI. GI cancer mortality in participants in low dose CT screening for lung cancer with a focus on pancreatic cancer. Sci Rep. 2024 Dec 2;14(1):29851. doi: 10.1038/s41598-024-76322-z. PMID 39617764